CLINICAL TRIAL: NCT05996471
Title: A Phase 2b Multicenter, Randomized, Open-Label Study Comparing the Efficacy, Safety, PK, and Tolerability of VH3810109, Administered Either Intravenously Or As A Subcutaneous Infusion With rHuPH20, in Combination With CAB LA to Standard of Care in Virologically Suppressed Adults Living With HIV
Brief Title: A Study to Investigate the Virologic Efficacy and Safety of VH3810109 + Cabotegravir Compared to Standard of Care (SOC) in Male and Female Adults Living With Human Immunodeficiency Virus (HIV)
Acronym: EMBRACE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 209639
Record Dates: First submitted 2023-08-09; First posted 2023-08-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections
Keywords: VH3810109; Cabotegravir; Standard of care; HIV; Long acting; Virologically Suppressed
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Part 1A: Participants Receiving VH3810109 Formulation 1 plus Cabotegravir (Experimental): Participants will receive VH3810109 formulation 1 intravenously (IV) and Cabotegravir intramuscularly (IM) every month (QM). Participants from this arm will either transition to Part 2A or discontinue from the study and enter the LTFU period.
  Interventions: Biological: VH3810109; Drug: Cabotegravir
- Part 1B: Participants Receiving VH3810109 plus rHuPH20 plus Cabotegravir (Experimental): Participants will receive VH3810109 plus rHuPH20 via subcutaneous (SC) infusion and Cabotegravir IM. This arm was discontinued following preliminary results. Participants from this arm will either transition to Part 1A at the next dosing visit or withdraw from the Investigational Product (IP) and enter the LTFU.
  Interventions: Biological: VH3810109; Drug: Cabotegravir; Biological: rHuPH20
- Part 1C: Participants Receiving SOC ART (Active Comparator): Participants in this arm will either transition to Part 2B or Part 2C or discontinue from the study.
  Interventions: Drug: Standard of care (SOC)
- Part 2A: Participants Receiving VH3810109 Formulation 2 plus Cabotegravir Q2M (Experimental): Participants will receive VH3810109 formulation 2 intravenously (IV) and Cabotegravir intramuscularly (IM) every 2 months (Q2M). Participants from this arm will either transition to Part 3A or discontinue from the study and enter the LTFU period.
  Interventions: Biological: VH3810109; Drug: Cabotegravir
- Part 2B: Participants Receiving VH3810109 Formulation 2 plus Cabotegravir (Experimental): Participants will receive VH3810109 formulation 2 intravenously (IV) and Cabotegravir intramuscularly (IM) at Day 1, Month 1, Month 2 and then Q2M. Participants from this arm will either transition to Part 3A or discontinue from the study and enter the LTFU period.
  Interventions: Biological: VH3810109; Drug: Cabotegravir
- Part 2C: Participants continuing SOC ART (Active Comparator): Participants in this arm will either transition to Part 3B or discontinue from the study.
  Interventions: Drug: Standard of care (SOC)
- Part 3A: Participants continuing VH3810109 Formulation 2 plus Cabotegravir Q2M (Experimental): Participants will continue to receive VH3810109 formulation 2 intravenously (IV) and Cabotegravir intramuscularly (IM) every 2 months (Q2M).
  Interventions: Biological: VH3810109; Drug: Cabotegravir
- Part 3B: Participants receiving VH3810109 Formulation 2 plus Cabotegravir (Experimental): Participants will receive VH3810109 formulation 2 intravenously (IV) and Cabotegravir intramuscularly (IM) at Day 1, Month 1, Month 2 and then Q2M.
  Interventions: Biological: VH3810109; Drug: Cabotegravir

INTERVENTIONS:
Biological: VH3810109 — VH3810109 will be administered.
  Arms: Part 1A: Participants Receiving VH3810109 Formulation 1 plus Cabotegravir; Part 1B: Participants Receiving VH3810109 plus rHuPH20 plus Cabotegravir; Part 2A: Participants Receiving VH3810109 Formulation 2 plus Cabotegravir Q2M; Part 2B: Participants Receiving VH3810109 Formulation 2 plus Cabotegravir; Part 3A: Participants continuing VH3810109 Formulation 2 plus Cabotegravir Q2M; Part 3B: Participants receiving VH3810109 Formulation 2 plus Cabotegravir
Drug: Cabotegravir — Cabotegravir will be administered.
  Arms: Part 1A: Participants Receiving VH3810109 Formulation 1 plus Cabotegravir; Part 1B: Participants Receiving VH3810109 plus rHuPH20 plus Cabotegravir; Part 2A: Participants Receiving VH3810109 Formulation 2 plus Cabotegravir Q2M; Part 2B: Participants Receiving VH3810109 Formulation 2 plus Cabotegravir; Part 3A: Participants continuing VH3810109 Formulation 2 plus Cabotegravir Q2M; Part 3B: Participants receiving VH3810109 Formulation 2 plus Cabotegravir
Drug: Standard of care (SOC) — Pre-baseline SOC antiretroviral therapy (ART) will be administered.
  Arms: Part 1C: Participants Receiving SOC ART; Part 2C: Participants continuing SOC ART
Biological: rHuPH20 — rHuPH20 will be administered.
  Arms: Part 1B: Participants Receiving VH3810109 plus rHuPH20 plus Cabotegravir

SUMMARY:
The study aims at evaluating the efficacy of VH3810109, dosed in accordance with the dosing schedule as either intravenous (IV) infusion or subcutaneous (SC) infusion with recombinant hyaluronidase (rHuPH20), in combination with cabotegravir (CAB) intramuscular (IM) dosed in accordance with the dosing schedule in virologically suppressed, Antiretroviral therapy (ART)-experienced adult participants living with HIV. VH3810109 plus rHuPH20 plus Cabotegravir arm of the study has been discontinued based on preliminary results. The study will be conducted in 3 parts followed by a Long-Term Follow-up phase (LTFU).

ELIGIBILITY:
Inclusion criteria

Age

1. Participant must be 18 to 70 years of age inclusive, at the time of signing the informed consent.

   Type of Participant and Disease Characteristics
2. Must be on uninterrupted current regimen for at least 6 months prior to Screening. Any prior switch, defined as a change of a single drug or multiple drugs simultaneously, must have occurred due to tolerability/safety, access to medications, or convenience/simplification, and must NOT have been done for treatment failure (HIV-1 RNA ≥200 c/mL).

   Acceptable stable - ARV regimens prior to Screening include at least one NRTI plus:
   * INSTI
   * NNRTI
   * Boosted PI (or atazanavir [ATV] unboosted)
   * Excludes current use of cabotegravir or fostemsavir

   The addition, removal, or switch of a drug(s) that has been used to treat HIV based on antiretroviral properties of the drug constitutes a change in ART with the following limited exceptions:
   * Historical changes in formulations of ART drugs or booster drugs will not constitute a change in ART regimen if the data support similar exposures and efficacy, and the change must have been at least 3 months prior to Screening.
   * Historical maternal perinatal use of an NRTI when given in addition to an ongoing HAART will not be considered a change in ART regimen.
   * A change in dosing scheme of the same drug from twice daily to once daily will not be considered a change in ART regimen if data support similar exposures and efficacy.

   For Part 2

   • Any participant who has received or is currently receiving an INSTI at the time of screening must be on their first INSTI-containing regimen and must not have used any other INSTIs previously
3. Documented evidence of at least two plasma HIV-1 RNA measurements <50 c/mL in the 12 months prior to Screening: one within the 6 to 12-month window, and one within 6 months prior to Screening;
4. Plasma HIV-1 RNA <50 c/mL at Screening;
5. Screening CD4+ T-cell count ≥350 cells/mm3:

   Weight
6. Body weight >=50 kg to <=115 kg.

   Sex
7. Male and/or female Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies, assuring minimal contraception requirements noted below.

All participants participating in the study should be counselled on safer sexual practices including the use and benefit/risk of effective barrier methods (e.g. male condom) and on the risk of HIV transmission to an uninfected partner.

1. Participants who are female at birth are eligible to participate if at least one of the following conditions applies:

   * Not pregnant or breastfeeding and at least one of the following conditions applies:

     * Is not a participant of childbearing potential (POCBP). OR
     * Is a POCBP and using an acceptable contraceptive method during the intervention period (at a minimum until after the last dose of study intervention). The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.
   * A POCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) on Day 1, prior to the first dose of study intervention.

     * If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
   * The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a POCBP with an early undetected pregnancy.

   QTc 8. QTc Interval <450 msec.

   Phenotypic Sensitivity 9. Viral phenotypic sensitivity to VH3810109 based on IC90 of <=2 ug/mL and a Maximum Percent Inhibition >98% using the Monogram PhenoSense mAb Assay on sample obtained at a screening visit.

   Informed Consent 10. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

   Exclusion Criteria:

   Medical conditions:

   • Participants who are pregnant, breastfeeding, plan to become pregnant or breastfeed during the study
   * Participants having skin disease or disorder (i.e. infection, inflammation, dermatitis, eczema, drug rash, drug allergy, psoriasis, food allergy, urticaria) or tattoo overlying potential injection sites which may interfere with interpretation of injection site reactions or administration of VH3810109 or CAB
   * Participant has a gluteal implant/enhancement (including fillers) overlying the gluteus area or any other area which may significantly interfere with interpretation of injection site reactions
   * Participants with known history of cirrhosis with or without viral hepatitis co-infection
   * Participants with ongoing or clinically relevant pancreatitis
   * Untreated syphilis infection (positive rapid plasma reagin (RPR) at screening) without documentation of treatment. Participants who are at least 7 days post completed treatment are eligible if recruitment is open
   * Prior receipt of licensed or investigational HIV monoclonal antibody
   * Any evidence of an active Centers for Disease Control and Prevention (CDC) Stage 3 disease except cutaneous Kaposi's sarcoma not requiring systemic therapy. Historical or current CD4 cell counts less than 200 cells/mm^3 are not exclusionary
   * History of sensitivity to any of the study medications or their components or drugs of their class, or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation
   * Any condition which, in the opinion of the investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs, cART or render the participant unable to take oral medication
   * Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening
   * Previous exposure to cabotegravir
   * Participant enrolled in a prior or concurrent clinical study that includes a drug intervention within the last 30 days
   * Participants with chronic hepatitis B (HBsAg positive) infection
   * Individuals who are co-infected with HIV and Hepatitis B virus (HBV) will be excluded.
   * Participants with hepatitis C co-infection
   * Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
   * Participants who in the investigator's judgment, pose a significant suicidality risk
   * Contraindications, as per the current Prescribing Information for cabotegravir.
   * Previous hypersensitivity reaction to cabotegravir or
   * Contraindicated co-administered drugs:

     * Anticonvulsants: Carbamazepine, oxcarbazepine, phenobarbital, phenytoin
     * Antimycobacterials: Rifabutin, rifampin, rifapentine
     * Glucocorticoid (systemic): Dexamethasone (more than a single-dose treatment)
     * Herbal product: St John's wort (Hypericum perforatum)

   Prior/Concomitant Therapy:

   • Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.

   • Previous exposure to cabotegravir.
   * Treatment with any of the following agents within 60 days of screening:

     -radiation therapy;
     * cytotoxic chemotherapeutic agents;
     * any systemic immune suppressant.
   * Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of study medication.
   * Current or anticipated need for chronic anti-coagulants.
   * Participants receiving any prohibited medication and who are unwilling or unable to switch to an alternate medication.

   Prior/Concurrent Clinical Study Experience • Participant enrolled in a prior or concurrent clinical study that includes a drug intervention within the last 30 days.

   Diagnostic Assessments • Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the participants inclusion in the study of an investigational compound.

   • Any evidence of viral resistance based on the presence of any major cabotegravir resistance-associated mutation [IAS-USA, 2022] in any historic resistance test result.
   * Any verified Grade 4 laboratory abnormality with the exception of Grade 4 triglycerides or lipid abnormalities. A single repeat test is allowed during the Screening period to verify a result.
   * Alanine aminotransferase (ALT) >=3 times the upper limit of normal (ULN)
   * Creatinine clearance of <50 mL/min/1.73 m^2 via using the refitted, race-neutral Chronic Kidney Disease Epidemiology Collaboration (CKD-EPIcr_R) method.
   * PT >=Grade 2 (>=1.25 ULN). A single repeat test is allowed during the Screening period to verify a result.

   Other Exclusion Criteria

   • To assess any potential impact on participant eligibility with regard to safety, the investigator must refer to the IB and supplements, approved product labels, and/or local prescribing information for detailed information regarding warnings, precautions, contraindications, AEs, drug interactions, and other significant data pertaining to the study drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2028-11-09 (Estimated)

PRIMARY OUTCOMES:
Part 1 and Part 2B and 2C: Number of Participants with Plasma HIV-1 Ribonucleic acid (RNA) Greater Than or Equal to (≥)50 Copies per Millilitre (c/mL) per Snapshot Algorithm at Month 6 | Month 6

SECONDARY OUTCOMES:
Part 1, 2 and 3: Number of Participants with Serious Adverse Events (SAEs), Deaths, and Adverse Events (AEs) Leading to Discontinuation of Investigational Product (IP) | Up to Month 24
Part 1, 2 and 3: Number of Participants with Grade 3-4 AEs | Up to Month 24
Part 1, 2 and 3: Number of Participants with Grade 3-4 Laboratory Abnormalities | Up to Month 24
Part 1, 2 and 3: Number of Participants with Grade 1-4 Injection/infusion Site Reactions | Up to Month 24
Part 1, 2 and 3: Number of Participants Meeting Confirmed Virologic Failure (CVF) Criteria over time | Up to Month 24
Part 1, 2 and 3: Number of Participants with Plasma HIV-1 RNA ≥50 c/mL per Snapshot Algorithm Over Time | Up to Month 24
Part 1, 2 and 3: Number of Participants with Plasma HIV-1 RNA Less Than (<)50 c/mL per Snapshot Algorithm Over Time | Up to Month 24
Part 1, 2 and 3: Number of Participants with HIV Disease Progression | Up to Month 24
Part 1, 2 and 3: Serum Concentrations of VH3810109 | Up to Month 24
Part 1, 2 and 3: Plasma Concentrations of Cabotegravir | Up to Month 24
Part 1, 2 and 3: Absolute Value for Cluster of Differentiation 4 (CD4+) T-Cell Count | Up to Month 24
Part 1, 2 and 3: Change from Baseline in CD4+ T-Cell Count | Baseline (Day 1) and up to Month 24
Part 1, 2 and 3: Absolute Value for Cluster of Differentiation 8 (CD8+) T-Cell Count | Up to Month 24
Part 1, 2 and 3: Change from Baseline in CD8+ T-Cell Count | Baseline (Day 1) up to Month 24
Part 1, 2 and 3: Number of Participants with Anti-VH3810109 Antibodies | Up to Month 24
Part 1, 2 and 3: Number of Participants with Neutralizing Antibodies Against VH3810109 | Up to Month 24
Part 1, 2 and 3: Number of Participants with Treatment-emergent Genotypic Resistance | Up to Month 24
Part 1, 2 and 3: Number of Participants with Treatment-emergent Phenotypic Resistance | Up to Month 24

CONTACTS AND LOCATIONS:
Locations (39):
- United States (38):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Southfield, Michigan
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Watertown, Wisconsin
- GSK Investigational Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/